CLINICAL TRIAL: NCT06883695
Title: A Phase Ⅰ, Randomized, Double-Blind, Placebo-Controlled Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-3045 in Healthy Subjects
Brief Title: A Phase Ⅰ Clinical Trial to Evaluate the Safety, Tolerance, Pharmacokinetics and Pharmacodynamics of SHR-3045 in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-3045-101
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-3045 Group (Experimental)
  Interventions: Drug: SHR-3045 Injection
- SHR-3045 Placebo Group (Placebo Comparator)
  Interventions: Drug: SHR-3045 Placebo Injection

INTERVENTIONS:
Drug: SHR-3045 Injection — SHR-3045 injection.
  Arms: SHR-3045 Group
Drug: SHR-3045 Placebo Injection — SHR-3045 placebo injection.
  Arms: SHR-3045 Placebo Group

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR-3045 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with ability to understand the trial procedures and possible adverse events, voluntary participation in the trial.
2. Subjects who can provide written informed consent.
3. Males or females aged 18-55 years (both inclusive).
4. Males with body weight ≥ 50 kg, or females with body weight ≥ 45 kg.
5. No clinically significant abnormalities in the medical history, general physical examinations, vital signs and laboratory tests.

Exclusion Criteria:

1. Participation in clinical trials of other investigational drugs or medical devices within 3 months prior to screening.
2. Known or suspected history of drug abuse.
3. Addiction to tobacco and alcohol.
4. Individuals who are unable to adhere to the dietary requirements of this trial during the study period.
5. Judged by the investigator, there are any other conditions that interfere with the results evaluation of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | From screening period up to day 113.

SECONDARY OUTCOMES:
Area under the concentration-time curve from time 0 to the last time point after SHR-3045 administration (AUC0-last). | Post-dose at day 1 to day 113.
Area under the concentration-time curve from time 0 to infinity after SHR-3045 administration (AUC0-inf). | Post-dose at day 1 to day 113.
Maximum observed concentration of SHR-3045 (Cmax). | Post-dose at day 1 to day 113.
Time to maximum observed concentration of SHR-3045 (Tmax). | Post-dose at day 1 to day 113.
Clearance of SHR-3045 (CL). | Post-dose at day 1 to day 113.
Terminal elimination half-life of SHR-3045 (t1/2). | Post-dose at day 1 to day 113.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided